CLINICAL TRIAL: NCT00939588
Title: An 8 Week, Double-blind, Randomized, Parallel-group Study to Compare the Effect of Aliskiren 300mg + Valsartan 320mg vs. Telmisartan 80mg + Ramipril 10mg on Biomarkers of the Renin-angiotensin-aldosterone System in Moderate Hypertension
Brief Title: Compare the Effect of Aliskiren Plus Valsartan Versus Angiotensin-Converting Enzyme Inhibitor (ACEi) Plus Angiotensin Receptor Blocker (ARB) [Ramipril Plus Telmisartan] on the Renin-Angiotensin-Aldosterone System (RAAS) in Hypertensive Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CSPV100A2225
Record Dates: First submitted 2009-07-09; First posted 2009-07-15 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Hypertension
Keywords: Aliskiren,; hypertension,; renin-angiotensin-aldosterone system
MeSH Terms: conditions — Hypertension | interventions — aliskiren; Valsartan; Telmisartan; Ramipril

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Aliskiren and Valsartan (Experimental)
  Interventions: Drug: Aliskiren/ Valsartan
- Telmisartan and Ramipril (Active Comparator)
  Interventions: Drug: Telmisartan/ Ramipril

INTERVENTIONS:
Drug: Aliskiren/ Valsartan
  Arms: Aliskiren and Valsartan
Drug: Telmisartan/ Ramipril
  Arms: Telmisartan and Ramipril

SUMMARY:
This study is designed as a mechanistic study to compare the effect of two different combinations of anti-hypertensive treatments (aliskiren and valsartan vs. telmisartan and ramipril) on the renin-angiotensin-aldosterone system (RAAS) in patients with moderate hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Males or females of non-childbearing potential, 18 to 65 years of age with moderate hypertension
* Patients who are eligible and able to participate in the study

Exclusion criteria:

* Severe hypertension or secondary form of hypertension.
* Serum potassium > 5.1 mEq/L (mmol/L)
* Heart failure
* Any history of hypertensive encephalopathy or cerebrovascular accident; any history of TIA, myocardial infarction, coronary bypass surgery or percutaneous coronary intervention
* Uncontrolled or life-threatening arrythmia

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-07; Primary Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Compare the effects of aliskiren + valsartan vs ramipril + telmisartan on 24-hour urinary aldosterone | 56 days

SECONDARY OUTCOMES:
Compare the effects of aliskiren + valsartan vs ramipril + telmisartan on Plasma Renin Activity (PRA)and angiotensin II | 56 days
Compare the effects of aliskiren + valsartan vs ramipril + telmisartan on mean sitting systolic and diastolic blood pressure | 56 days
Assess safety and tolerability of aliskiren + valsartan and ramipril + telmisartan | 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, Moscow, Russia